CLINICAL TRIAL: NCT06444685
Title: Motor and Cognitive Effects of Table Tennis on Parkinson's Disease: Pilot Controlled Trial
Brief Title: Effects of Table Tennis for People With Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Collaborators: Club Tennis Taula Borges Blanques (Unknown); Asociació de Parkinson de les Terres de Lleida (Unknown)
Responsible Party: Principal Investigator, Helena Fernández-Lago, Lecturer, Universitat de Lleida
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023CRINDESTABC
Record Dates: First submitted 2024-03-12; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Table Tennis (Experimental): Participants will follow supervised Table Tennis sessions lasting 60 minutes during 6 weeks, for a total of 12 sessions.
  Interventions: Other: Exercise and cognitive training interventino
- Tabletop Games (Experimental): Participants will follow supervised Tabletop Game sessions lasting 60 minutes during 6 weeks, for a total of 12 sessions.
  Interventions: Other: Exercise and cognitive training interventino

INTERVENTIONS:
Other: Exercise and cognitive training interventino — Exercise and cognitive training based on Table tennis and Tabletop games.

SUMMARY:
Quasi-experimental, controlled, non-randomised two-arm pilot, with an experimental group (table tennis exercise) and an active control group (cognitive training based on board games).

DETAILED DESCRIPTION:
Quasi-experimental, controlled, non-randomised two-arm pilot, with an experimental group (table tennis exercise) and an active control group (cognitive training based on board games). Interventions in both groups will take place twice a week for 6 weeks (12 sessions in total). The main variables to be assessed will be motor and cognitive. As secondary variables, clinical and daily life aspects will be assessed. As results, it is expected that the experimental group will obtain improvements in motor variables compared to the control group after receiving the interventions. However, improvements in cognitive variables and secondary variables are expected to be similar in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease based on the UK PD Society Brain Bank Criteria
* Stage I to III on the Hoehn and Yahr scale
* Ability to walk for 10 minutes unassisted

Exclusion Criteria:

* Score of under 23 on the Mini-Mental State Examination
* Severe Visual or Auditory deficits
* Cardiovascular conditions that impede physical activity
* Brain surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Amplitude of Center of Pressure under simple conditions | Assessed before starting the intervention (T0) and 6 weeks later (T0 + 6 weeks).
  Assessment of amplitude of Center of Pressure (in mm) during balance testing using OPAL Sensors (APDM, Oregon, USA).
Amplitude of Center of Pressure under Dual Task conditions (Motor) | Assessed before starting the intervention (T0) and 6 weeks later (T0 + 6 weeks).
  Assessment of amplitude of Center of Pressure (in mm) during balance testing under concurrent cognitive tasks (Motor, by holding a glass of water on a tray) using OPAL Sensors (APDM, Oregon, USA).
Amplitude of Center of Pressure under Dual Task conditions (Arithmetic) | Assessed before starting the intervention (T0) and 6 weeks later (T0 + 6 weeks).
  Assessment of amplitude of Center of Pressure (in mm) during balance testing under concurrent cognitive tasks (Arithmetic, by concurrently substracting 7 from a random number) using OPAL Sensors (APDM, Oregon, USA).
Amplitude of Center of Pressure under Dual Task conditions (Verbal) | Assessed before starting the intervention (T0) and 6 weeks later (T0 + 6 weeks).
  Assessment of amplitude of Center of Pressure (in mm) during balance testing under concurrent cognitive tasks (Verbal, by naming words starting by a random letter) using OPAL Sensors (APDM, Oregon, USA).
Trail-Making Test | Assessed before starting the intervention (T0) and 6 weeks later (T0 + 6 weeks).
  Assessment of Trail-Making Test parts A and B

SECONDARY OUTCOMES:
United Parkinson's Disease Rating Scale - Part III | Assessed before starting the intervention (T0) and 6 weeks later (T0 + 6 weeks).
  Assessment of Motor symptoms of Parkinson's Disease with a predetermined assessment
Montreal Cognitive Assessment | Assessed before starting the intervention (T0) and 6 weeks later (T0 + 6 weeks).
  Assessment of cognitive status to detect Mild Cognitive Impairment with a preset questionnaire.
Parkinson's Disease Questionnaire - 8 | Assessed before starting the intervention (T0) and 6 weeks later (T0 + 6 weeks).
  Assessment of Quality of Life for people with Parkinson's Disease through a self-administered questionnaire
Timed Up and Go test | Assessed before starting the intervention (T0) and 6 weeks later (T0 + 6 weeks).
  Assessment of gait mobility and fall risk by getting up from a chair, walking 3 meters, turning back and sitting again.
Falls Efficacy Scale International | Assessed before starting the intervention (T0) and 6 weeks later (T0 + 6 weeks).
  Assessment of perceived fall risk with a predetermined questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recerca Biomèdica de Lleida, Lleida, Spain

REFERENCES:
- [Background] Alexander GE, Crutcher MD, DeLong MR. Basal ganglia-thalamocortical circuits: parallel substrates for motor, oculomotor, "prefrontal" and "limbic" functions. Prog Brain Res. 1990;85:119-46. PMID 2094891
- [Background] Shahed J, Jankovic J. Motor symptoms in Parkinson's disease. Handb Clin Neurol. 2007;83:329-42. doi: 10.1016/S0072-9752(07)83013-2. No abstract available. PMID 18808920
- [Background] Inoue K, Fujioka S, Nagaki K, Suenaga M, Kimura K, Yonekura Y, Yamaguchi Y, Kitano K, Imamura R, Uehara Y, Kikuchi H, Matsunaga Y, Tsuboi Y. Table tennis for patients with Parkinson's disease: A single-center, prospective pilot study. Clin Park Relat Disord. 2020 Dec 30;4:100086. doi: 10.1016/j.prdoa.2020.100086. eCollection 2021. PMID 34316664
- [Background] Olsson K, Franzen E, Johansson A. A Pilot Study of the Feasibility and Effects of Table Tennis Training in Parkinson Disease. Arch Rehabil Res Clin Transl. 2020 Jun 2;2(3):100064. doi: 10.1016/j.arrct.2020.100064. eCollection 2020 Sep. PMID 33543090
- [Background] Estrada-Plana V, Montanera R, Ibarz-Estruga A, March-Llanes J, Vita-Barrull N, Guzman N, Ros-Morente A, Ayesa Arriola R, Moya-Higueras J. Cognitive training with modern board and card games in healthy older adults: two randomized controlled trials. Int J Geriatr Psychiatry. 2021 Jun;36(6):839-850. doi: 10.1002/gps.5484. Epub 2021 Jan 8. PMID 33275804